CLINICAL TRIAL: NCT01917903
Title: The Effects of Dual Task Treadmill Training on Gait and Cognition in Individuals With Parkinson's Disease.
Brief Title: Cognitive-motor Training for PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Lisa Muratori, Associate Professor, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 64249
Record Dates: First submitted 2013-07-30; First posted 2013-08-07 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Parkinson's Disease
Keywords: walking; Parkinson's disease; physical therapy; falls; memory; attention; multitasking; exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Assessments are performed by a clinician blinded to participant group (training vs. waitlist control) allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Identification of at risk variables (Experimental): Individuals will come in for a single visit to perform all tasks / conditions. Measurements will be taken of spatial and temporal features of walking with and without a secondary task. In addition, cognitive tests of memory and attention will be performed. Outcomes will narrow measures to those most likely to show clinically significant change.
  Interventions: Behavioral: Identification of at risk variables
- Gait-Cognitive training (Experimental): Participants will engage in a four week treadmill training program with a secondary cognitive component aimed at improving both walking and multitasking.
  Interventions: Behavioral: Gait-cognitive training

INTERVENTIONS:
Behavioral: Gait-cognitive training — Participants will engage in a four week treadmill training program with a secondary cognitive component aimed at improving both walking and multitasking.
  Arms: Gait-Cognitive training
Behavioral: Identification of at risk variables — Participants will complete walking under three conditions: walking alone for six minutes; standing from a chair, walking 3 meters, turning, and returning to a seated position (TUG); and standing from a chair, walking 3 meters turning and returning to a seated postion while subtracting numbers (TUG Cognitive). Spatiotemporal measures of gait will be collected.
  Arms: Identification of at risk variables

SUMMARY:
This study will evaluate gait when individuals with Parkinson's disease (PD) are walking and how walking changes when challenged to perform a functional cognitive task simultaneously. By looking at walking alone and walking with varying cognitive loads the investigators will be able to determine motor and cognitive factors vulnerable to interference in PD. Each is important to understand so that training can address components of walking that become impaired when someone is distracted by a common cognitive task and so that the intensity of treatment matches the level of task difficulty. Using this initial data, the investigators will establish a protocol to improve walking taking into account the unique features of PD, including bradykinesia, freezing of gait, stiffness, and problems with memory and attention. The investigators will evaluate the potential for this treatment to improve walking and improve or maintain cognitive abilities necessary to multitask.

DETAILED DESCRIPTION:
In this study participants will be asked to participate in a training study to examine whether a new walking intervention that combines cognitive training with walking on a treadmill improves walking more than gait training or cognitive training alone. Participants with Parkinson's disease (PD) will come to the lab for a complete gait assessment using a motion analysis system that will record leg motion and muscle activity during comfortable walking. During the initial evaluation, participants will also complete cognitive assessments and surveys about community activities and quality of life related to PD. Participants will be divided into two training groups and asked to come to the lab three times a week for four weeks during the intervention. One week and one month after training, participants will return to the lab to complete all the same assessments that were performed during the initial visit. The results of the three testing sessions (initial, one week and one month) will be compared between and within groups to see if any of the interventions provided unique benefits to the health of persons with PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease with our without cognitive impairment
* ambulatory for at least 200 feet without an assistive device (cane, walker, etc)

Exclusion Criteria:

* recent orthopedic injury (e.g., fracture, sprain, muscle pull, herniated disc)
* concurrent neurological illnesses including stroke, brain cancer, spinal cord injury, and diabetic neuropathies.
* cardiac insufficiency limiting ability to participate in walking study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Spatiotemporal measures of gait across conditions and over time. | Baseline testing at day one of study; follow-up testing at three time periods: 4-5 weeks after baseline (immediate post-training); 5-6 weeks (one week post-training); and 9-10 weeks after baseline (one month post-training)
  Changes in gait parameters are a key measure of the difficulty of performing two tasks at once. Decreases in gait speed, increased time in double support (two feet on the ground) and stopping while talking have been linked to increased disability and risk for falls.

SECONDARY OUTCOMES:
Changes in cognitive performance measured with serial sevens. | Baseline (day one); week 4-5 (immediate post 4 week training program); 5-6 weeks (one-week post-training); 9-10 weeks (one month post-training)
  Participants will count backward by sevens from a digit between 90 and 100. The ability to perform the task will be used as a measure of cognitive trade-off relative to walking performance.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Muratori, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University RRAMP Laboratory, Stony Brook, New York, United States